CLINICAL TRIAL: NCT02770105
Title: Neurophysiological Correlates of L-theanine, Caffeine and Their Combination on Improving Selective Attention in a Visual Reaction Time Task: A Functional Magnetic Resonance Imaging (fMRI) Study
Brief Title: Theanine and Caffeine on Neurophysiology of Attention
Acronym: THECNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Single
Other Study IDs: TTUIRB505445
Record Dates: First submitted 2016-05-06; First posted 2016-05-12 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-05

CONDITIONS: L-theanine
Keywords: L-theanine; caffeine; selective attention; fMRI; RVRT
MeSH Terms: interventions — theanine; Caffeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Theanine — Oral administration of 200mg of L-theanine powder dissolved in 200ml of distilled water
Other: Caffeine — Oral administration of 160mg of anhydrous caffeine powder dissolved in 200ml of distilled water
Other: Theanine-Caffeine Combination — Oral administration of 200mg of L-theanine and 160mg of anhydrous caffeine powder, dissolved in 200ml of distilled water
Other: Placebo — Oral administration of 200ml of distilled water

SUMMARY:
L-theanine and caffeine are nutritional compounds that are naturally found in tea. Our recent findings using an EEG paradigm are consistent with the findings of others, indicating that intake of L-theanine and caffeine reduce the time needed for a person to differentiate between two visual stimuli and react to only one stimulus. In order to understand how these compounds give rise to these improvements, the investigators need to study how these compounds are related to various areas of the brain. To achieve this, the investigators plan to scan the brains of nine participants after they take either 1) L-theanine alone, 2) caffeine alone 3) the combination of both L-theanine and caffeine as compared with a placebo (distilled water), to see which has the greatest impact on attention and on regions in the brain that bring about attention.

DETAILED DESCRIPTION:
Recruitment: Participants will be recruited through advertisements in social media, electronic and hardcopy noticeboards at Texas Tech University (e.g. Tech Announce, campus bulletin boards), local media (e.g. newspapers), web-based media (e.g. Craig's list) and flyers placed on bulletin boards off campus. Nine participants will be recruited after screening for the following inclusion and exclusion criteria.

Pre-Screening (Telephone): Individuals who express an interest in participating will be contacted by a graduate or an undergraduate research assistant who will administer a structured telephone interview to: 1) provide information related to the requirements of the study, along with potential risks and benefits 2) Screen for eligibility based on specific inclusion and exclusion criteria. All potential subjects will be informed that their responses will remain confidential and that taking part in the screening interview in no way obligates them to participate.

The first 9 participants who meet eligibility criteria will be scheduled for their appointments (at Texas Tech Neuroimaging Institute; TTNI) immediately or within 48 hours of the telephone conversation depending on the discretion of each potential participant. Each participant will be required to complete 5 visits to TTNI, scheduled at least 5 days apart, in order to complete their participation in the study. The first visit will be 45 minutes in length and each of the 4 subsequent visits will be 90 minutes in length. The participants will be given the right to withdraw from the study at any point. In the event that a screened and included participant should discontinue the study prematurely, additional subjects will be recruited to maintain study total at 9 completers. Since the study is a cross-over design, all participants will be exposed to all experimental conditions (i.e. theanine, caffeine, TC and distilled water) in a random order.

Measurements:

1. Recognition Visual Reaction Time (RVRT) Task: Participants will be instructed on the importance of accuracy in performing the RVRT task in advance. A blue-colored background will be presented. Participants will be requested to press a button on a computer keyboard (during practice sessions) and on a fiber optic hand-held device during active testing sessions (in the fMRI scanner) using the index finger of the dominant hand in response to a white flash lasting for 30ms (target stimulus) as quickly as possible, while ignoring a red colored flash lasting for 30ms (distractor stimulus). During each run, 20±2 stimuli of each category of stimuli will be presented and the inter-stimulus interval will be jittered to 5000ms±3000ms. Time taken to respond to target stimuli will be recorded as RVRT. Omissions and responses to distractor stimuli (errors) will also be recorded.
2. Scanning paradigm: Each scanning session will be scheduled for 20 minutes, comprised of 3 runs of fMRI scans while the participants are performing the RVRT tasks displayed on an LCD screen and projected via a mirror attached to the head coil of the fMRI machine (each run lasting for 4 minutes) followed by a structural (T1-weighted) scan lasting for 5 minutes.

Data Collection Protocol: All recruited participants will be scheduled for 5 visits at the TTNI within 48 hours of receipt and subsequent evaluation of the prescreening material for inclusion and exclusion criteria. Participants will be reminded of the visits via email / telephone (per their stated preference) at both 1 week and again 1 day prior to each visit. The visits will be scheduled at least 5 days apart.

1. First Visit: Prescreening, Consent and Training:

   1. The study will be explained thoroughly to reinforce prior explanations and ensure full understanding.
   2. Participants will be screened again to verify the inclusion and exclusion criteria by re-administering the screening questionnaire and MRI safety sheet by a member of the BMTR lab.
   3. Informed written consent will be obtained.
   4. A participant number will be assigned, that identifies the order of administration of the four substances (i.e. theanine, caffeine, TC and placebo) during the subsequent visits. This order will be determined using a random number generator.
   5. Each participant will be provided with a solution of 160mg of caffeine dissolved in 200ml of distilled water in a disposable, clean, opaque, plastic cup to be consumed completely within 1 minute, in order to train the participants to consume required substances during the subsequent visits and to ensure that the participants can tolerate the mildly bitter taste of the substances.
   6. In order to acclimate the participants to the RVRT task they will be performing in the MRI scanner during their subsequent visits, each participant will perform a training session where they will perform the RVRT task in three 5 min sessions, separated by 60 second rest intervals using a laptop computer (under the supervision of a graduate / undergraduate research assistants).
   7. Each participant will be reminded of the subsequent visits and the importance of adherence to the preparation guidelines.
2. Preparation and Administration of Substances: L-theanine and caffeine will be purchased in purified powder form from a registered supplier. Both substances will be stored in air-tight packing prior to preparation for administration according to manufacturer's recommendations. All solutions will be prepared for administration maintaining the highest possible standards of hygiene. Each solution of L-theanine will be made by dissolving 200mg of theanine powder in 200ml of distilled water. Each solution of caffeine will be made by dissolving 160mg of caffeine powder. Both L-theanine and caffeine powder (200mg and 160mg respectively) will be dissolved in a 200ml aliquot of distilled water to form each solution of TC. Two-hundred milliliters of distilled water will be used as the placebo. Each solution will be prepared within 4 hours of scheduled time of administration and stored in a disposable, clean, opaque, cup with a lid. The participants will be instructed to consume the solution completely upon administration.
3. Preparation of participants for the Second, Third, Fourth and Fifth Visits: All recruited participants will be instructed to strictly adhere to the following guidelines prior to the 2nd, 3rd, 4th and 5th visits in order to minimize confounding of the results.

   1. Avoid consumption of alcohol within 48 hours prior to the test
   2. Avoid smoking 12 hours prior to the test
   3. Sleep for at least 6 hours on the day prior to the test dates
   4. Avoid consumption of tea, coffee or foods / beverages containing caffeine within 12 hours prior to the test.
4. Second, Third, Fourth and Fifth Visits: Administration of Substances and MRI Scanning:

   1. Participants will be briefly reminded of the purpose of the study.
   2. Adherence to the preparation guidelines will be assessed. Should a participant indicate non-adherence to preparation guidelines they will be discontinued from the study.
   3. The solution (containing the appropriate substance / combination of substances) to be administered to each participant during the visit will be provided in a disposable, clean, cup to be consumed within 1 minute.
   4. A questionnaire regarding the taste and characteristics of the solution will be administered.
   5. Each participant will be given a verbal review of the RVRT task and will be allowed to practice the RVRT task on a laptop computer for 5 minutes.
   6. Each participant will be allowed to relax, seated in a comfortable chair, until 60 minutes elapses from the time of administration of the solution (to allow time for the actions of L-theanine and caffeine on the brain to reach the maximum levels).
   7. Combined functional and structural MRI scans will be performed while the participants engage in the RVRT tasks.
   8. Visual analogue scales (100mm lines with the extremes of the measured parameter listed at each end; the participant rates the measured parameter by making a vertical mark on the line) will be administered to measure the perceived improvement / deterioration of RVRT and perceived improvement / deterioration of accuracy in the tasks
   9. At the end of the 5th visit, each participant will be debriefed.

Analysis: RVRT will be compared across the four conditions (theanine, caffeine, TC and placebo) constructing a repeated measures analysis of variance (ANOVA) model using the R-statistical software. Subsequently, pair-wise comparisons of RVRT will be performed between the four conditions, maintaining the family-wise error rate at 0.05. Following sequence of operations will be conducted on the fMRI data using the FMRIB software library (FSL): visual examination, distortion correction, motion correction, slice timing correction, spatial smoothing and statistical analysis. BOLD responses will be compared across the four conditions by constructing ANOVA models at a whole brain level as well as in the regions of anterior cingulate cortex and antero-medial prefrontal cortex. Pair-wise comparisons of BOLD responses will also be conducted between the conditions. RVRT, omissions and errors will be included as covariates in fMRI analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males*
* Age 18-60 years

Exclusion Criteria:

* Gross impairment of vision or hearing that would prevent the participants from recognizing visual stimuli
* Physical, psychiatric or neurological impairment that could affect cognitive or motor functions
* Exposure to toxins or substances that are known to affect visual, auditory, cognitive or motor functions
* Regular intake of medication that could alter visual, auditory, cognitive or motor functions
* History of and / or current alcohol and / or drug abuse
* Disease or condition known to be precipitated or aggravated by tea or coffee
* Intake of drugs containing caffeine, other phosphodiesterase inhibitors or adenosine receptor blockers
* Intake of medications which are known to have pharmacological interactions with caffeine
* Participants with contra-indications to undergo fMRI scanning
* Unwilling or unable to discontinue the use of cell phones, smart phones or other electronic devices during the entire study visit.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Differences between fMRI blood oxygen level dependent (BOLD) responses of the brain recorded following administration of each substance and the placebo | Sixty minutes after administration of each of theanine, caffeine, theanine-caffeine combination and placebo
  Theanine, caffeine, theanine-caffeine combination and distilled water (placebo) will be administered on 4 separate days (at least 5 days apart) in a random order. Functional MRI scans will be performed 60 minutes after each administration. Primary outcome measure will be the difference in fMRI BOLD responses obtained for each substance and the placebo.

SECONDARY OUTCOMES:
Differences between mean recognition visual reaction times recorded following administration of each substance and the placebo | Sixty minutes after administration of each of theanine, caffeine, theanine-caffeine combination and placebo
  Theanine, caffeine, theanine-caffeine combination and distilled water (placebo) will be administered on 4 separate days (at least 5 days apart) in a random order. Functional MRI scans will be performed 60 minutes after each administration. A secondary outcome measure will be the difference in mean recognition visual reaction time task obtained for each substance and the placebo, when the subjects perform the task in the fMRI scanner.
Differences between proportion of errors caused while performing the recognition visual reaction time task following administration of each substance and the placebo | Sixty minutes after administration of each of theanine, caffeine, theanine-caffeine combination and placebo
  Theanine, caffeine, theanine-caffeine combination and distilled water (placebo) will be administered on 4 separate days (at least 5 days apart) in a random order. Functional MRI scans will be performed 60 minutes after each administration. A secondary outcome measure will be the difference in proportion of errors caused while performing the recognition visual reaction time task in the fMRI scanner after each substance and the placebo.
Differences between proportion of omissions caused while performing the recognition visual reaction time task following administration of each substance and the placebo | Sixty minutes after administration of each of theanine, caffeine, theanine-caffeine combination and placebo
  Theanine, caffeine, theanine-caffeine combination and distilled water (placebo) will be administered on 4 separate days (at least 5 days apart) in a random order. Functional MRI scans will be performed 60 minutes after each administration. A secondary outcome measure will be the difference in proportion of omissions caused while performing the recognition visual reaction time task in the fMRI scanner after each substance and the placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Binks, PhD, Principal Investigator — Texas Tech University - Department of Nutritional Sciences
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahathuduwa CN, Dassanayake TL, Amarakoon AMT, Weerasinghe VS. Acute effects of theanine, caffeine and theanine-caffeine combination on attention. Nutr Neurosci. 2017 Jul;20(6):369-377. doi: 10.1080/1028415X.2016.1144845. Epub 2016 Feb 12. PMID 26869148
- [Background] Weerasinghe V, Kahathuduwa C, Amarakoon T, Dassanayake T. Synergistic Effect of Theanine and Caffeine on Visual Reaction Time, Evoked Potentials and Cognitive Event Related Potentials. Journal of Clinical Neurophysiology. 2015; 32(4): S396.
- [Background] Camfield DA, Stough C, Farrimond J, Scholey AB. Acute effects of tea constituents L-theanine, caffeine, and epigallocatechin gallate on cognitive function and mood: a systematic review and meta-analysis. Nutr Rev. 2014 Aug;72(8):507-22. doi: 10.1111/nure.12120. Epub 2014 Jun 19. PMID 24946991